CLINICAL TRIAL: NCT04466956
Title: Virtual Reality as a Distraction Technique for the Management of Acute Pain and Anxiety During Manual Vacuum Aspiration for Miscarriage
Brief Title: Virtual Reality in MVA for Miscarriage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: North Middlesex University Hospital NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 271029
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Miscarriage
Keywords: Management; Anxiety; Pain
MeSH Terms: conditions — Abortion, Spontaneous; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Intervention 25 and control 25
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality for reduction of pain and anxiety during MVA (Active Comparator): 25 participants randomised to use VR headset during MVA and complete questionnaire and short interview regarding experience
  Interventions: Device: Virtual reality
- Control group- no VR (No Intervention): 25 participants randomised to not use VR headset during MVA and complete questionnaire and short interview regarding experience

INTERVENTIONS:
Device: Virtual reality — Virtual reality headset worn with short relaxing video played during MVA procedure
  Arms: Virtual reality for reduction of pain and anxiety during MVA

SUMMARY:
We are investigating the use of a virtual reality programme to reduce pain and anxiety experienced during manual vacuum aspiration.

Virtual reality (VR) is the computer-generated simulation of a three-dimensional environment that can be interacted with in a seemingly real way by a person using special electronic equipment. In this study a VR headset is worn by the patient allowing them to experience a relaxing environment whilst the procedure manual vacuum aspiration (MVA) is performed.

VR is mostly used in computer gaming but has uses in medical field and has been used in the treatment of long standing pain, treatment of burns, dentistry and treatment of cancer pain. However, its role in the management of pain and anxiety during gynaecological procedures like manual vacuum aspiration has not been researched. This study explores whether it has a place in the treatment of gynaecological pain and reduction of anxiety.

DETAILED DESCRIPTION:
Many simple gynaecological procedures can be performed in an outpatient setting without the need for general anaesthesia. Such office-based procedures include outpatient hysteroscopy, endometrial biopsy, large-loop-excision of the transformation zone and manual vacuum aspiration for the management of miscarriage. Advantages experienced by patients include reduced anaesthetic risk, enhanced recovery time and flexibility of timings. For the healthcare provider there are significant cost benefits on the basis of reduced theatre time, staff and equipment. Patient satisfaction is generally high but influenced by their experience of pain and feelings of anxiety before, during and after the procedure.

The rationale for this study is to invetsigate the role of distraction techniques and the feasibility of using virtual reality for the management of acute pain and anxiety experienced by patients undergoing manual vacuum aspiration

Primary objective

• Feasibility of using virtual reality as a distraction technique in management of acute pain and anxiety in patients undergoing manual vacuum aspiration for miscarriage.

Secondary objectives

* Understanding the acceptability and effectiveness of VR interventions in office gynaecology procedures
* Understanding the factors that might influence the willingness of patients to participate in a future formal trial of the technology.
* Understanding how best to implement the technology and designing of the contents of the VR intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients: Clinical indications for undergoing an MVA will be confirmed. Inclusion criteria will include all women of 18 - 50 years of age, planned for a MVA who are able and willing to give informed consent.

Exclusion Criteria:

* Hearing impairments and blindness
* History of epilepsy or any previous seizures
* Any known anatomical characteristics that may make performing the office procedure more difficult (e.g., cervical conisation)
* Any known characteristics that make the patient unsuitable for undergoing MVA (e.g. known bleeding disorder, gestation >12 weeks)
* The denial or withdrawal of informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nandita Deo, MRCOG, Principal Investigator — Barts & The London NHS Trust
Locations (2):
- United Kingdom (2):
  - Whipps Cross University Hospital, London
  - North Middlesex University Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At completion of study anticipated 2022
Access Criteria: Public

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2021- July 2022 across 2 sites: Whipps Cross University Hospital (WCUH) and North Middlesex University Hospital (NMUH).
  Consecutive women with retained products of pregnancy post miscarriage or abortion attending emergency gynaecology/early pregnancy units at both sites were offered inclusion if they fulfilled inclusion criteria.
Pre-assignment Details: In both participating hospitals, MVAs are offered as an option for management of missed or incomplete miscarriage, or retained pregnancy tissue after abortion. Eligibility criteria included patients aged 18 - 50 years who were able to give written, informed consent. Patients were excluded if they were unable to speak fluent English; had hearing or visual impairments; or a history of epileptic seizures or claustrophobia
Period: Overall Study
Arm/Group | Virtual Reality for Reduction of Pain and Anxiety During MVA | Control Group- no VR
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 50 patients agreed to participate from the 72 eligible women approached and offered inclusion
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality for Reduction of Pain and Anxiety During MVA | Control Group- no VR | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (6.9) | 33 (5.1) | 32.5 (6.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 25 | 25 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weeks gestation [Mean (Standard Deviation); unit: weeks] | 9.3 (2.1) | 9.0 (2.1) | 9.15 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Rating
Description: Anxiety score (numerical rating score 0 least-10 worst) and questionnaire
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality for Reduction of Pain and Anxiety During MVA | Control Group- no VR
Number analyzed (Participants) | 25 | 25
score on a scale | 4.4 (3.2) | 3.94 (2.4)

2. Primary Outcome: Pain Rating
Description: Pain score (numerical rating score 0 least-10 worst) and questionnaire
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality for Reduction of Pain and Anxiety During MVA | Control Group- no VR
Number analyzed (Participants) | 25 | 25
score on a scale | 5.54 (2.2) | 4.68 (2.3)
Statistical Analysis 1: Comparison: Virtual Reality for Reduction of Pain and Anxiety During MVA vs Control Group- no VR; Mean worst pain scores were 5.98 and 6.88 in the standard care and VR groups respectively, with difference in means -0.9 (95% CI -2.1 - 0.28), p value 0.13. Mean anxiety scores at the end of the procedure were 3.94 and 4.4 in the standard care and VR groups respectively, with difference in means -0.46 (95% CI -2.1, 1.1), p value 0.57; Test type: Other — Statistical analysis was by intention-to-treat including all randomised participants, using Stata-12 software. Continuous data were summarised as mean and standard deviation, and categorical data as counts and percentages. Between group differences were reported with 95% confidence intervals, and p-values, using t-test to compare normally distributed data and chi-squared tests to compare categorical data; p < 0.01, t-test, 1 sided — Between group differences were reported with 95% confidence intervals, and p-values, using t-test to compare normally distributed data and chi-squared tests to compare categorical data

ADVERSE EVENTS:
Time Frame: 1 year (July 2021-July 2022)
Description: No adverse events occurred
Arm/Group | Virtual Reality for Reduction of Pain and Anxiety During MVA | Control Group- no VR
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04466956/Prot_SAP_000.pdf